CLINICAL TRIAL: NCT02895009
Title: A Randomized Comparison of TR Band Hemostatic Compression Patterns After Transradial Coronary Intervention
Brief Title: Hemostatic Compression Patterns After Transradial Coronary Intervention
Acronym: HCPATRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016yzdh19
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; Radial artery occlusion; transradial coronary intervention
MeSH Terms: conditions — Coronary Disease; Arterial Occlusive Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Other): Participants allocated to the control group will receive a routine long term postoperative puncture site compression via TR Band. In control group, TR Band deflation is commenced at the 2nd hour with successive 5 mL air released at 2 hours intervals until the bladder was empty at the 6th hour, and the TR Band is removed at the 24th hour.
  Interventions: Device: control group
- experimental group (Experimental): Participants allocated to the experimental group will receive a short term postoperative puncture site compression via TR Band. In experimental group, TR Band deflation is commenced at the 1st hour with 3 mL air released, and at the 2nd hour with 5ml, and at the 3rd hour with the remainder air in the bladder, and the TR Band is removed at the 12th hour.
  Interventions: Device: experimental group

INTERVENTIONS:
Device: experimental group — Participants allocated to the experimental group will receive a short term postoperative puncture site compression via TR Band. TR Band deflation is commenced at the 1st hour and completed at the 3rd hour, and the TR Band is removed at the 12th hour.
  Arms: experimental group
Device: control group — Participants allocated to the control group will receive a routine long term postoperative puncture site compression via TR Band. TR Band deflation is commenced at the 2nd hour and completed at the 6th hour, and the TR Band is removed at the 24th hour.
  Arms: control group

SUMMARY:
The purpose of the study is to investigate the protective effects of short term TR Band compression on transradial coronary occlusion after transradial coronary intervention.

DETAILED DESCRIPTION:
Radial artery occlusion (RAO), an infrequent but serious complication after transradial coronary intervention (TRI), prevents subsequent use of the same radial artery for coronary angiography and intervention. Comparing to the overseas counterparts, most Chinese medical workers put more emphasis on prevention of postoperative puncture site bleeding, so longer compression hemostasis time is applied but this prolonged compression may underestimate or even ignore an increasing risk of RAO. Therefore, this study intends to compare short term TR Band compression and the routine long term one on transradial coronary occlusion after transradial coronary intervention.

Participants allocated to the control group will receive a routine long term postoperative puncture site compression via TR Band. In control group, TR Band deflation is commenced at the 2nd hour with successive 5 mL air released at 2 hours intervals until the bladder was empty at the 6th hour, and the TR Band is removed at the 24th hour.

Participants allocated to the experimental group will receive a short term postoperative puncture site compression via TR Band. In experimental group, TR Band deflation is commenced at the 1st hour with 3 mL air released, and at the 2nd hour with 5ml, and at the 3rd hour with the remainder air in the bladder, and the TR Band is removed at the 12th hour.

At the 24th hour, RAO incidence, postoperative puncture site bleeding incidence and patient comfort level will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patients who received TRI for the first time

Exclusion Criteria:

* Failure to puncture the radial artery in 1 attempt
* Inaccessible radial arteries because of anatomic variations, such as hypoplastic radial arteries and radioulnar loop, which can be confirmed by radial artery angiography before the TRI
* Patients who had previous radial procedure
* Patients who were receiving IIb/IIIa receptor antagonist treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
RAO incidence | at the 24th hour post TRI
  At the 24th hour post TRI, RAO will be diagnosed via ultrasonic sound and RAO incidence will be evaluated between two groups.

SECONDARY OUTCOMES:
postoperative puncture site bleeding incidence | within 24 hours after TRI
  postoperative puncture site bleeding incidence will be studied in patient between two groups within 24 hours after TRI.
patient comfort level | at the 24th hour post TRI
  At the 24th hour post TRI, patient comfort level will be evaluated by patients via a visual analogue scale for comfort level.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Hu, Master, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

REFERENCES:
- [Background] Campeau L. Percutaneous radial artery approach for coronary angiography. Cathet Cardiovasc Diagn. 1989 Jan;16(1):3-7. doi: 10.1002/ccd.1810160103. PMID 2912567
- [Background] Kiemeneij F, Laarman GJ. Percutaneous transradial artery approach for coronary stent implantation. Cathet Cardiovasc Diagn. 1993 Oct;30(2):173-8. doi: 10.1002/ccd.1810300220. PMID 8221875
- [Background] Rathore S, Stables RH, Pauriah M, Hakeem A, Mills JD, Palmer ND, Perry RA, Morris JL. A randomized comparison of TR band and radistop hemostatic compression devices after transradial coronary intervention. Catheter Cardiovasc Interv. 2010 Nov 1;76(5):660-7. doi: 10.1002/ccd.22615. PMID 20506228
- [Background] Dai N, Xu DC, Hou L, Peng WH, Wei YD, Xu YW. A comparison of 2 devices for radial artery hemostasis after transradial coronary intervention. J Cardiovasc Nurs. 2015 May-Jun;30(3):192-6. doi: 10.1097/JCN.0000000000000115. PMID 24496325
- [Background] Cong X, Huang Z, Wu J, Wang J, Wen F, Fang L, Fan M, Liang C. Randomized Comparison of 3 Hemostasis Techniques After Transradial Coronary Intervention. J Cardiovasc Nurs. 2016 Sep-Oct;31(5):445-51. doi: 10.1097/JCN.0000000000000268. PMID 26002786
- [Background] Fech JC, Welsh R, Hegadoren K, Norris CM. Caring for the radial artery post-angiogram: a pilot study on a comparison of three methods of compression. Eur J Cardiovasc Nurs. 2012 Mar;11(1):44-50. doi: 10.1177/1474515111429656. Epub 2012 Jan 11. PMID 22357780
- [Background] Pancholy SB, Patel TM. Effect of duration of hemostatic compression on radial artery occlusion after transradial access. Catheter Cardiovasc Interv. 2012 Jan 1;79(1):78-81. doi: 10.1002/ccd.22963. Epub 2011 May 16. PMID 21584923